CLINICAL TRIAL: NCT04292314
Title: Impact of Combination Therapy Between Hydroxy Urea, Omega 3, Nigella Sativa and Honey on Antioxidant-oxidant Status and Reduction of Iron Overload in Pediatric Major Thalassemia
Brief Title: Hydroxy Urea, Omega 3, Nigella Sativa,Honey on Oxidative Stress and Iron Chelation in Pediatric Major Thalassemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Maternity and Children Hospital, Makkah (Other); Beni-Suef Health insurance hospital (Unknown); University of Arizona (Other)
Responsible Party: Principal Investigator, Mohamed Medhat Abdelwahab Gamaleldin, Dr.Mohamed Medhat Abdelwahab Gamaleldin, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TQ/Omega-3 on Thalassemia
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Iron Overload; Oxidative Stress; Thalassemia Major
Keywords: thymoquinone; omega3; hydroxyurea; pediatric Thalassemia Major; oxidative stress; iron chelation; iron overload; chelation activity of thymoquinone; antioxidant effect of omega3; anti-hemolysis effect of hydroxyurea
MeSH Terms: conditions — Iron Overload; beta-Thalassemia | interventions — Docosahexaenoic Acids; Nigella sativa oil; Hydroxyurea; Honey; Deferoxamine

STUDY DESIGN:
Intervention Model Description: Four experimental groups, one control group.
  Each experimental group receives different experimental treatments plus traditional treatment in the hospital and the control group receives only traditional treatment.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Omega-3 experimental group (Experimental): 50 patients from each participating hospital that will receive Omega-3 supplementation (300-400mg EPA & 200-300mg DHA) per day for 8 consecutive months up to 10 months.
  in addition to experimental treatment this group will receive the traditional treatment of deferoxamine/deferasirox plus regular blood transfusion with dose de-escalation methods till efficacy of experimental treatment proved.
  Interventions: Drug: Omega 3; Drug: Deferoxamine; Procedure: blood transfusion session
- Nigella sativa experimental group (Experimental): 50 patients from each participating hospital that will receive Nigella sativa supplementation (1g black seed oil contain 1% thymoquinone) per day for 8 consecutive months up to 10 months.
  in addition to experimental treatment this group will receive the traditional treatment of deferoxamine/deferasirox plus regular blood transfusion with dose de-escalation methods till efficacy of experimental treatment proved.
  Interventions: Drug: Nigella Sativa Oil; Drug: Deferoxamine; Procedure: blood transfusion session
- Hydroxyurea experimental group (Experimental): 50 patients from each participating hospital that will receive hydroxyurea medication (5 to 15mg/kg) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of deferoxamine/deferasirox plus regular blood transfusion with dose de-escalation methods until the efficacy of experimental treatment proved.
  Interventions: Drug: Hydroxyurea; Drug: Deferoxamine; Procedure: blood transfusion session
- Natural honey experimental group (Experimental): 50 patients from each participating hospital that will receive natural honey(2.5 mg/kg dissolved in 250 ml water) per day for 8 consecutive months up to 10 months.
  in addition to the experimental treatment, this group will receive the traditional treatment of deferoxamine/deferasirox plus regular blood transfusion with dose de-escalation methods until the efficacy of experimental treatment proved.
  Interventions: Drug: Honey; Drug: Deferoxamine; Procedure: blood transfusion session
- Ordinary hospital treatment group (Active Comparator): 50 patients from each participating hospital that will receive the ordinary treatment of iron chelator agent of deferoxamine or deferasirox (SubQ infusion: 20 to 40 mg/kg/day over 8 to 12 hours, 6 to 7 nights per week, maximum daily dose: 40 mg/kg/day)for 8 consecutive months up to 10 months.
  in addition to iron chelator agent, this group receive regular blood transfusion session.
  Interventions: Drug: Deferoxamine; Procedure: blood transfusion session

INTERVENTIONS:
Drug: Omega 3 — Omega-3 supplementation (300-400mg EPA & 200-300mg DHA) per day for 8 consecutive months up to 10 months
  Arms: Omega-3 experimental group
Drug: Nigella Sativa Oil — Nigella sativa supplementation (1g black seed oil contain 1% thymoquinone) per day for 8 consecutive months up to 10 months
  Arms: Nigella sativa experimental group
Drug: Hydroxyurea — hydroxyurea medication (5 to 15mg/kg) per day for 8 consecutive months up to 10 months.
  Arms: Hydroxyurea experimental group
Drug: Honey — Natural honey(2.5 mg/kg dissolved in 250 ml water) per day for 8 consecutive months up to 10 months.
  Other Names: Natural honey formulation
  Arms: Natural honey experimental group
Drug: Deferoxamine — deferoxamine (SubQ infusion: 20 to 40 mg/kg/day over 8 to 12 hours, 6 to 7 nights per week, maximum daily dose: 40 mg/kg/day)for 8 consecutive months up to 10 months.
Procedure: blood transfusion session — Regular blood transfusion session based on patient hematological profile starts from one session every 2 weeks.

SUMMARY:
The aim of the present study is evaluating the strength of combination therapy of hydroxy urea, omega 3, nigella sativa and honey on antioxidant-oxidant status (OXIDATIVE STRESS) in response to reactive oxygen species production (LIPID PEROXIDATION) and their effect on iron intoxication (IRON CHELATION) in pediatric major thalassemia.

DETAILED DESCRIPTION:
Beta thalassemia is a blood disorder that reduces the production of hemoglobin. Hemoglobin is the iron-containing protein in red blood cells that carries oxygen to cells throughout the body. In people with beta thalassemia, low levels of hemoglobin lead to a lack of oxygen in many parts of the body. Affected individuals also have a shortage of red blood cells (anemia), which can cause pale skin, weakness, fatigue, and more serious complications. People with beta thalassemia are at an increased risk of developing abnormal blood clots. Beta thalassemia is classified into two types depending on the severity of symptoms: thalassemia major (also known as Cooley's anemia) and thalassemia intermedia. Of the two types, thalassemia major is more severe.

Beta-thalassemia syndromes are a group of hereditary blood disorders. It is characterized by reduced beta globin chain synthesis, resulting in reduced Hb in red blood cells (RBC), decreased RBC production and anemia.

Homozygotes for beta-thalassemia may develop either thalassemia major or thalassemia intermedia. Individuals with thalassemia major usually come to medical attention within the first 2 years and require regular blood transfusion to survive.

Affected infants with thalassemia major fail to thrive and become progressively pale. Feeding problems, diarrhea, irritability, recurrent bouts of fever, and enlargement of the abdomen, caused by splenomegaly, may occur. If a regular transfusion program that maintains a minimum Hb concentration of 95-105 g/L is initiated, then growth and development are normal until the age of 10-11 years. After the age of 10-11 years, affected individuals are at risk of developing severe complications related to posttransfusional iron overload, depending on their compliance with chelation therapy.

Complications of iron overload include growth retardation and failure of sexual maturation and also those complications observed in adults with hemachromatosis -associated hereditary hemochromatosis (HH): involvement of the heart (dilated myocardiopathy and pericarditis), liver (chronic hepatitis, fibrosis, and cirrhosis), and endocrine glands (resulting in diabetes mellitus and insufficiency of the parathyroid, thyroid, pituitary, and, less commonly, adrenal glands).

The underlying basis of b-thalassemia pathology is the diminished b-globin synthesis leading to a-globin accumulation and premature apoptotic destruction of erythroblasts, causing oxidative stress-induced ineffective erythropoiesis.

ELIGIBILITY:
Inclusion Criteria:

1. Any case with full manifestation of β-THALASSEMIA major disease
2. #Aged from 7-15 years old
3. # accompanied with ineffective erythropoiesis
4. # with low hemoglobin level
5. # with iron overload

Exclusion Criteria:

1. The presence of any other chronic illness.
2. Patient age>15 years old or < 7 years old.
3. The presence of concomitant myocardial infarction, stroke, acute chest syndrome.
4. The patient suffers from any other type of anemia.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
F 2 -isoprostanes pg/mL | 3 months
  plasma F 2 -isoprostanes Picograms Per Millilitre measured by high pressure liquid chromatography assay
Total cholesterol Mg/dl | 10 months
  Total cholesterol milligrams per deciliter
HDL cholesterol Mg/dl | 10 months
  HDL cholesterol milligrams per deciliter
LDL cholesterol Mg/dl | 10 months
  LDL cholesterol milligrams per deciliter
Triglycerides Mg/dl | 10 months
  Triglycerides milligrams per deciliter
Serum total iron mcg/dL | 10 months
  Serum total iron micrograms per decilitre
% transferrin saturation | 10 months
  transferrin saturation percentage
C-reactive protein mg/L | 10 months
  C-reactive protein milligrams per deciliter
Serum Ferritin ng/ml | 10 months
  Serum Ferritin Nanograms per milliliter
Total Iron Binding Capacity (TIBC) mcg/dL | 10 months
  Total Iron Binding Capacity micrograms per decilitre
hemoglobin (Hbg) g/dL | 10 months
  hemoglobin (Hbg) gram/deciliter
mean corpuscular hemoglobin (MCH) pg/ml | 10 months
  mean corpuscular hemoglobin (MCH) Picograms Per Millilitre
leukocytes count μl | 10 months
  leukocytes in microliter
% Chelation activity Fe+++ - thymoquinone complex | 3 months
  Chelation activity of Ferric - thymoquinone complex in percentage measured by high pressure liquid chromatography coupled with gaschromatography - mass spectroscopy analysis
% Chelation activity Fe++ - thymoquinone complex | 3 months
  Chelation activity of Ferrous - thymoquinone complex in percentage measured by high pressure liquid chromatography coupled with gaschromatography- mass spectroscopy analysis
Lactic acid dehydrogenase U/L | 10 months
  Lactic acid dehydrogenase unit per litter
Reticulocyte count % | 10 months
  Reticulocyte count percentage
Hb-F level g/dL | 10 months
  hemoglobin- F level in gram per deciliter
Reticulocyte absolute count | 10 months
  Reticulocyte absolute count in a cubic milliliter of blood
White blood cells count | 10 months
  White blood cells count in a cubic milliliter of blood

CONTACTS AND LOCATIONS:
Overall Officials: IVO IBRAHAM [Prof of Pharmacy, Clinical Translational Sciences], Ph.D., Study Director — University of Arizona, College of Pharmacy; AHMED A ALBERRY [Assistant prof of clinical pharmacology], Ph.D., Study Director — Beni-Suef University, Faculty of medicine; RAGHDA R SAYED [Lecturer of Clinical Pharmacy], Ph.D., Study Director — Beni-Suef University, Faculty of Pharmacy; MOHAMED M ABDELWAHAB GAMALELDIN, Ph.D Student, Principal Investigator — Beni-Suef University, Faculty of Pharmacy; Mohamed H Meabad [Prof of Pediatrics], M.D, Study Director — Beni-Suef university, Faculty of medicine; Ahmed F Mahmoud Hussein, MS.c, Study Director — Beni-Suef Health insurance hospital
Locations (4):
- Egypt (3):
  - Faculty of medicine, Beni-suef univeristy - Beni-Suef university hospital, Banī Suwayf
  - Faculty of Pharmacy, Beni-Suef university, Banī Suwayf
  - Health insurance hospital, Banī Suwayf
- Maternity and Children hospital, Mecca, Saudi Arabia